CLINICAL TRIAL: NCT02938208
Title: An Investigation to Test a Prototype Full-face Mask in the Home Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-198
Record Dates: First submitted 2016-10-16; First posted 2016-10-19 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Jupiter Full Face Mask (Experimental): Participants to use full face mask in-home for a 14 ± 3 days in-home.
  Interventions: Device: Jupiter Full Face Mask

INTERVENTIONS:
Device: Jupiter Full Face Mask — Full Face Mask for the treatment of obstructive sleep apnea (OSA) using CPAP therapy.

SUMMARY:
This investigation is a prospective non-blinded and non-randomized clinical investigation. This investigation is designed to evaluate the performance (leak and comfort) as well as participant's overall acceptance of the Jupiter mask amongst OSA participants. A total number of up to 15 OSA participants who currently use full face masks will be recruited for the trial.

DETAILED DESCRIPTION:
This investigation is designed to evaluate the performance (leak and comfort) as well as participant's overall acceptance of the Jupiter mask amongst OSA participants. A total number of up to 15 OSA participants who currently use full face masks will be recruited for the trial. The participants will be recruited from the Fisher and Paykel Healthcare Database of subjects with OSA (Ethics reference NTY/08/06/064), Auckland District Health Board (ADHB), or WellSleep Centre (Bowen Hospital, Wellington, NZ).

Participants will be on the trial for 21 days ± 6 days, using the prototypes at home for 14 days ± 3 days. PAP baseline data on the participant's prescribed treatment pressure with their usual mask and will be collected for 7 days ± 3 days prior to mask fitting with the Jupiter trial mask.

Fisher and Paykel Healthcare will act as the investigator and sponsor for this investigation. This study will be conducted in accordance with ICH/GCP Guidelines. No deviation from the protocol will be implemented without prior review and approval of the sponsor except where it may be necessary to eliminate an immediate hazard to a research participant. In such case, the deviation will be reported to the sponsor (Bhavi Ogra) as soon as possible.

ELIGIBILITY:
Inclusion Criteria

* 18+ years of age
* Diagnosed with OSA by a practicing physician
* Prescribed PAP therapy (Bi-Level or Continuous Positive Airway Pressure (CPAP) or Automatic Positive Airway Pressure (APAP)). Patient can be naïve to CPAP therapy or experienced (6 months and more)
* Existing full face mask users
* Patients who are able to put on and remove their current mask without gross difficulty relating to an existing condition (e.g. arthritis of the hands).

Exclusion Criteria

* Inability to give informed consent
* Anatomical or physiological conditions making PAP therapy inappropriate (e.g unconsolidated facial fracture)
* Commercial Drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or think they may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Objective mask leak data measurement (System Leak) | Up to 21 ± 6 days in-home
  Obtained from participant's CPAP device, measured in L/min
Subjective Measurement of leak assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire
Comfort assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire
Stability assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire
Draft assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire
Noise assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire

SECONDARY OUTCOMES:
Preference of Mask assessed using a Subjective Questionnaire | Up to 21 ± 6 days in-home
  Subjective Questionnaire
Usability via mask unboxing/fitting exercise with a subjective questionnaire | Up to 21 ± 6 days in-home
  Usability activity during visit 2 with subjective questionnaire after activity

CONTACTS AND LOCATIONS:
Overall Officials: Kayan Gonda, BSc, Principal Investigator — Sponsor Employee
Locations (2):
- New Zealand (2):
  - Fisher & Paykel Healthcare, Auckland
  - Wellsleep: Bowen Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No
This is an investigation for a prototype full face mask. The results from this trial will feedback into product development on further improving the full face mask for future trials and impending release of the product.